CLINICAL TRIAL: NCT03759288
Title: A 52-Week, Multicenter, Randomized, Double-blind, Placebo and Active-Controlled, Operationally Seamless Phase 2b/3, Parallel-group Study to Assess the Efficacy and Safety of Brazikumab in Participants With Moderately to Severely Active Crohn's Disease (INTREPID Lead-In)
Brief Title: An Active and Placebo-Controlled Study of Brazikumab in Participants With Moderately to Severely Active Crohn's Disease
Acronym: INTREPID
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Strategic decision to discontinue the development of brazikumab in inflammatory bowel disease.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5271C00001; #3150-301-008 (Other: Legacy - Allergan); 2018-004346-42 (EudraCT Number)
Record Dates: First submitted 2018-11-20; First posted 2018-11-29 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-10

CONDITIONS: Crohn's Disease; IBD
Keywords: Crohn's Disease; Inflammatory bowel disease; Brazikumab; IL23 receptor; IBD; CD
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- (Stage 1) Brazikumab high dose (Experimental): Intravenous Brazikumab on Days 1, 29, and 57, followed by subcutaneous Brazikumab on Day 85 and every 4 weeks through Week 48
  Interventions: Drug: Brazikumab high dose
- (Stage 1) Brazikumab low dose (Experimental): Intravenous Brazikumab on Days 1, 29, and 57, followed by subcutaneous Brazikumab on Day 85 and every 4 weeks through Week 48
  Interventions: Drug: Brazikumab low dose
- (Stage 1) Placebo (Placebo Comparator): Intravenous placebo on Days 1, 29, and 57, followed by subcutaneous placebo on Day 85 and every 4 weeks through Week 48
  Interventions: Drug: Placebo
- (Stage 2) Brazikumab high dose (Experimental): Intravenous Brazikumab on Days 1, 29, and 57, followed by subcutaneous Brazikumab on Day 85 and every 4 weeks through Week 48
  Interventions: Drug: Brazikumab high dose
- (Stage 2) Brazikumab low dose (Experimental): Intravenous Brazikumab on Days 1, 29, and 57, followed by subcutaneous on Day 85 and every 4 weeks through Week 48
  Interventions: Drug: Brazikumab low dose
- (Stage 2) Humira® (Active Comparator): Administered subcutaneously on Day 1, Day 15, and Day 29 and every 2 weeks through Week 50
  Interventions: Drug: Humira®

INTERVENTIONS:
Drug: Brazikumab low dose — Intravenous Brazikumab on Days 1, 29, and 57, followed by subcutaneous Brazikumab on Day 85 and every 4 weeks through Week 48
  Arms: (Stage 1) Brazikumab low dose; (Stage 2) Brazikumab low dose
Drug: Brazikumab high dose — Intravenous Brazikumab on Days 1, 29, and 57, followed by subcutaneous Brazikumab on Day 85 and every 4 weeks through Week 48
  Arms: (Stage 1) Brazikumab high dose; (Stage 2) Brazikumab high dose
Drug: Humira® — Administered subcutaneously on Day 1, Day 15, and Day 29 and every 2 weeks through Week 50.
  Arms: (Stage 2) Humira®
Drug: Placebo — Intravenous placebo on Days 1, 29, 57 followed by subcutaneous placebo on Day 85 and every 4 weeks through Week 48
  Arms: (Stage 1) Placebo

SUMMARY:
This study seeks to evaluate the safety and efficacy of brazikumab versus placebo (Stage I) and versus an active comparator (Stage 2) in participants with moderately to severely active CD and will include assessments of clinical response as demonstrated by improvement of symptoms and colonic mucosal appearance as observed on endoscopy

ELIGIBILITY:
Inclusion and Exclusion Criteria are the same for both Stage 1 and Stage 2; however, participants enrolled in Stage 1 will not be permitted to enroll in Stage 2.

Inclusion Criteria:

1. At the time of signing the informed consent, the participant must be 18 to 80 years of age, inclusive.
2. A diagnosis of ileal, ileocolonic, or colonic CD with an onset of symptoms for a minimum of 3 months prior to Screening as determined by the investigator based on clinical history, exclusion of other etiologies including infectious causes, and characteristic endoscopic and/or histologic findings.
3. Moderately to severely active CD defined by a CDAI score of 220 to 450 AND; CDAI LSF score ≥ 5 OR CDAI AP score ≥ 2; AND SES-CD of at least 6
4. Participant had an inadequate response or intolerance to intervention with conventional treatment [oral aminosalicylates, oral CS, azathioprine, methotrexate, or 6-mercaptopurine], or prior biological treatment, or demonstrated CS dependence for the treatment of CD. For participants who have previously used biological treatment, a participant may have failed up to 3 biologics that include up to 2 different mechanisms of action.
5. Participants taking 5-aminosalicylates, Oral prednisone (or equivalent), Budesonide, Immunomodulators, Oral antibiotics, Immunomodulators, Probiotics must be at a stable dose.
6. Participant must have the QFT-TB test performed and meet the following TB criteria.

A TB worksheet must also be completed:

1. Participant has no known history of active TB.
2. Participant has no known history of latent TB without completion of an appropriate course of intervention.
3. Meets 1 of the following acceptable TB test results:

i. Negative QFT-TB obtained from central laboratory during Screening, OR ii. For a positive QFT-TB test obtained during Screening from the central laboratory, active TB must be ruled out or treated and negative QFT-TB confirmed by central laboratory OR iii. Indeterminate QFT-TB test obtained during the Screening Period from the central laboratory with ongoing QFT-TB testing as outlined in Appendix G. Participants with an indeterminate QFT-TB test can continue with Screening if they have all of the following:

1. no symptoms/risk factors per TB worksheet provided by the sponsor
2. no known recent exposure to a case of active TB
3. no evidence of active TB on chest x-ray within 8 weeks prior to Screening or during Screening
4. confirmed QFT-TB negative by central laboratory

7 Female participants of childbearing potential must have a negative urine pregnancy test prior to administration of study intervention and must agree to use a highly effective method of birth control (confirmed by the investigator) from randomization throughout the study duration and for at least 18 weeks after last dose of study intervention.

8 Women not of childbearing potential are defined as women who are either permanently sterilized or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrhoeic for 12 months prior to the planned date of randomization without an alternative medical cause.

9 Nonsterilized males who are sexually active with a female partner of childbearing potential must comply with the methods of contraception during treatment and until the end of relevant systemic exposure in the male participant, plus a further 18 weeks.

10 Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.

11 Willingness and ability to attend all study visits, comply with the study procedures, read and write in order to complete questionnaires, and be able to complete the study period.

12 Provision of signed and dated written Optional Genetic Research Information informed consent prior to collection of samples for optional genetic research that supports Genomic Initiative.

Complete inclusion criteria are in the study protocol

Exclusion Criteria:

1. Participant is unable or unwilling to have endoscopic procedures performed during the study.
2. History or current diagnosis of ulcerative colitis, indeterminate colitis, microscopic colitis, ischemic colitis, colonic mucosal dysplasia, primary sclerosing cholangitis, or untreated bile acid malabsorption.
3. History of toxic megacolon within 3 months prior to Randomization.
4. Any intra-abdominal surgery, bowel resection, diversion, placement of ostomy or stoma within 3 months prior to Screening. Participants with a draining stoma, ostomy, or extensive colonic resection are excluded irrespective of the time from surgery.
5. Participant has an enterocutaneous or enterovesicular fistula. Participants with other active fistulas, including perianal fistulas, may be considered for enrollment if there is no anticipation for surgery and there is no evidence of active infection (eg, abscess).
6. Bowel perforation during the 6 months prior to Screening or evidence of obstruction within 3 months of Screening.
7. Complications of CD including short bowel syndrome, strictures/stenoses with obstruction or pre-stenotic dilation, or conditions where surgery may be anticipated within 6 months, or other conditions that may confound efficacy evaluations for the study.
8. Participant has any non-passable colonic stenosis/narrowing identified during the qualifying ileocolonoscopy (successful endoscope passage to the caecum with inability to enter the endoscope into the ileum is not covered under this exclusion criterion, and does not require exclusion).
9. Ongoing nutritional dependency for total parenteral nutrition or an elemental diet at Screening.
10. Participant has any of the following related to infections: • Evidence of a recent (within 6 months of Randomization) systemic fungal infection, requiring inpatient hospitalization, and/or antifungal treatment. • Any infection requiring hospitalization or treatment with IV anti-infectives (including antiviral treatment) within 4 weeks of Screening. • Cytomegalovirus or Epstein-Barr virus infection that has not resolved within 8 weeks prior to Screening • Clinically significant chronic infection (eg, osteomyelitis) that has not resolved within 8 weeks of Screening • Nonserious infection requiring oral anti-infectives within 2 weeks prior to randomization must be further discussed with the Study Physician/designee. • Participant has clinical evidence of or suspected to have an abscess during Screening. • Diagnosis of peritonitis or receiving treatment for peritonitis within 8 weeks prior to Screening • Participant has any underlying condition that predisposes participant to infections • Clinically significant active infection or signs/symptoms of infection that has the potential to worsen with immunosuppressive therapy • Signs or symptoms of ongoing infection due to intestinal pathogens
11. Previous allogenic bone marrow transplant or history of organ or cell-based transplantation (eg, islet cell transplantation or autologous stem cell transplantation) with the exception of corneal transplant.
12. Chronic hepatitis B or C infection.
13. Known history of primary immunodeficiency, splenectomy, or any underlying condition that predisposes the subject to infection, includingHIV infection.
14. Prior history of or current diagnosis of a demyelinating disorder.
15. Participant has received the following treatment: • Adalimumab, certolizumab pegol, infliximab, or golimumab: within 8 weeks prior to Randomization • Vedolizumab or ustekinumab within 12 weeks prior to Randomization • Other prohibited medication, biologic or small molecule treatment within 5 half-lives prior to Randomization • Fecal microbiota transplantation: within 8 weeks prior to Screening ileocolonoscopy
16. Except for ustekinumab, prior exposure to any biologic agent targeting IL-12 or IL-23.
17. Participants who received cyclosporine, mycophenolate mofetil, sirolimus (rapamycin), thalidomide, tacrolimus (FK-506), or tofacitinib within 2 weeks prior to Screening Visit 1.
18. Known history of allergy to the study intervention formulation or any of its excipients or components of the delivery device, or to any other biologic therapy.
19. Participants received more than 1 dose of IV or intramuscular steroids within 2 weeks prior to Screening Visit 1.
20. Participant received topical (rectal) aminosalicylic acid (eg, mesalamine) or topical (rectal) steroids within 2 weeks prior to Randomization.
21. Participant received a Bacille Calmette-Guérin vaccination within 12 months of Randomization or any other live vaccine less than 4 weeks prior to Randomization or is planning to receive any such vaccine over the course of the study.
22. Participant has known or suspected history of chronic use of NSAIDs (defined as at least 3 times per week for more than 3 months; not applicable to daily aspirin use up to 325mg per day) and/or opiates, drug, or alcohol abuse.
23. History of cancer with the following exceptions: (a) A history of basal cell carcinoma and/or squamous cell carcinoma of the skin, with apparent successful curative therapy greater than 12 months prior to Screening (b) Carcinoma in situ of the cervix, with apparent successful curative therapy, greater than 12 months prior to Screening.
24. Clinically significant cardiovascular conditions including recent myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, or Class III/IV heart failure within 6 months of Screening.
25. Prolonged QTcF interval (QTc >450 msec or QTC >480 for participants with bundle branch block; determined on central ECG), or conditions leading to additional risk for QT prolongation (eg, congenital long-QT syndrome).
26. Clinically significant kidney disease
27. Abnormal laboratory results at Screening
28. Other concurrent medical conditions: Participant has known, preexisting, clinically significant endocrine, autoimmune, metabolic, neurologic, renal, gastrointestinal, hepatic, hematological, respiratory or any other system abnormalities that are not associated with CD and are uncontrolled with standard treatment.
29. Participant is currently enrolled in another investigational device or drug study, or is within 35 days or 5 half-lives, whichever is longer, since ending another investigational device or drug study, or receiving other investigational agent(s)
30. Transfusion of blood, plasma, or platelets within the 30 days prior to Screening.
31. Females who are pregnant, nursing, or planning a pregnancy during the study OR females who are of childbearing potential and do not agree to use a highly effective method of contraception consistently and correctly.
32. Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals.
33. Previous randomization in the present study. . Complete exclusion criteria are in the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Stage 1. Percentage of patients with CDAI remission | at Week 12
  CDAI remission is defined as achieving the CDAI score below 150 (measured by PRO questionnaire and objective items (i.e. weight, hematocrit)).
Stage 2. Percentage of patients with endoscopic response | at Week 52
  Endoscopic response is described as minimum of 50% decrease from Baseline in SES-CD total score.
Stage 2. Percentage of patients with clinical remission | at Week 52
  Clinical remission is defined for a participant to satisfy the following two response thresholds simultaneously: average daily LSF subscore of ≤ 3 as assessed on the CDAI LSF item AND average daily AP subscore of ≤ 1 as assessed on the CDAI AP item (measured by PRO questionnaire).

SECONDARY OUTCOMES:
Stage 1. Percentage of patients with endoscopic response | at Week 12
  Endoscopic response is described as minimum of 50% decrease from Baseline in SES-CD total score.
Stage 1. Percentage of patients with clinical remission | at Week 12
  Clinical remission is defined for a participant to satisfy the following two response thresholds simultaneously: average daily LSF subscore of ≤ 3 as assessed on the CDAI LSF item AND average daily AP subscore of ≤ 1 as assessed on the CDAI AP item (measured by PRO questionnaire).
Stage 1. Percentage of patients with CDAI response | at Week 12
  CDAI response is defined as achieving the CDAI score of < 150 points or CDAI reduction from Baseline of ≥ 100 points (measured by PRO questionnaire and objective items (i.e. weight, hematocrit)).
Stage 1. Percentage of patients with CDAI remission | at both Week 12 and Week 52
  CDAI remission is defined as achieving the CDAI score below 150 (measured by PRO questionnaire and objective items (i.e. weight, hematocrit)).
Stage 1. Percentage of patients with CDAI response | at both Week 12 and Week 52
  CDAI response is defined as achieving the CDAI score of < 150 points or CDAI reduction from Baseline of ≥ 100 points (measured by PRO questionnaire and objective items (i.e. weight, hematocrit)).
Stage 1. Percentage of patients with endoscopic response | at both Week 12 and Week 52
  Endoscopic response is described as minimum of 50% decrease from Baseline in SES-CD total score.
Stage 1. Percentage of patients with clinical remission | at both Week 12 and Week 52
  Clinical remission is defined for a participant to satisfy the following two response thresholds simultaneously: average daily LSF subscore of ≤ 3 as assessed on the CDAI LSF item AND average daily AP subscore of ≤ 1 as assessed on the CDAI AP item (measured by PRO questionnaire).
Stage 1. Percentage of patients with endoscopic remission | at Week 52
  Endoscopic remission is defined as achieving the SES-CD total score of 0-2 OR SES-CD total score of ≤ 4 and at least 2 point reduction from Baseline with no subscore > 1
Stage 1. Percentage of patients with clinical remission | at Week 52
  Clinical remission is defined for a participant to satisfy the following two response thresholds simultaneously: average daily LSF subscore of ≤ 3 as assessed on the CDAI LSF item AND average daily AP subscore of ≤ 1 as assessed on the CDAI AP item (measured by PRO questionnaire).
Stage 1. Percentage of patients with CDAI response | at Week 52
  CDAI response is defined as achieving the CDAI score of < 150 points or CDAI reduction from Baseline of ≥ 100 points (measured by PRO questionnaire and objective items (i.e. weight, hematocrit)).
Stage 1. Percentage of patients with CDAI remission | at Week 52
  CDAI remission is defined as achieving the CDAI score below 150 (measured by PRO questionnaire and objective items (i.e. weight, hematocrit)).
Stage 1. Percentage of patients with endoscopic response | at Week 52
  Endoscopic response is described as minimum of 50% decrease from Baseline in SES-CD total score.
Stage 1. Percentage of patients with SES-CD total score of 0-2 | at Week 52
  SES-CD total score of 0-2
Stage 1. Percentage of patients with endoscopic response and endoscopic remission | Endoscopic response at Week 12, endoscopic remission at Week 52
  Endoscopic response: Minimum of 50% decrease from Baseline in SES-CD total score Endoscopic remission: SES-CD total score of 0-2, OR - SES-CD total score of ≤ 4 and at least 2 point reduction from Baseline with no subscore > 1
Stage 1. Serum concentration of brazikumab | Through Week 68
  Pharmacokinetics: concentration of brazikumab in serum
Stage 1. Incidence of anti-drug antibodies | Through Week 68
  Immunogenicity: incidence of brazikumab anti-drug antibodies in serum
Stage 1. Exposure-response | Through Week 68
  Derive exposure response model linking primary endpoint to metrics of model predicted individual brazikumab exposures
Stage 1. Serum IL-22 concentration clinical cutoff for Stage 2 | at Week 12
  Derive the relationship between baseline serum IL-22 concentration and efficacy of brazikumab through CDAI remission and endoscopic response
Stage 1. Number and percentage of patients with adverse events | Through Week 68
  Number and percentage of patients with reported adverse events.
Stage 1. Percentage of patients with potentially clinically significant changes in laboratory values | Through Week 68
  Percentage of patients with clinically significant changes in hematology, clinical chemistry, urinalysis.
Stage 1. Percentage of patients with potentially clinically significant changes in vital signs | Through Week 68
  Percentage of patients with potentially clinically significant changes in systolic, diastolic pulse rate.
Stage 1. Percentage of patients with potentially clinically significant changes in physical exams | Through Week 68
  Percentage of patients with potentially clinically significant changes in full physical exams.
Stage 1. Percentage of patients with potentially clinically significant changes in ECGs | Through Week 68
  Percentage of patients with potentially clinically significant changes in 12-lead ECG recordings
Stage 2. Percentage of patients with endoscopic response | at both Week 12 and Week 52
  Endoscopic response is described as minimum of 50% decrease from Baseline in SES-CD total score
Stage 2. Percentage of patients with clinical remission | at both Week 12 and Week 52
  Clinical remission is defined for a participant to satisfy the following two response thresholds simultaneously: average daily LSF subscore of ≤ 3 as assessed on the CDAI LSF item AND average daily AP subscore of ≤ 1 as assessed on the CDAI AP item (measured by PRO questrionare)
Stage 2: Percentage of patients with endoscopic remission | at Week 52
  Endoscopic remission: - SES-CD total score of 0-2, OR - SES-CD total score of ≤ 4 and at least 2 point reduction from Baseline with no subscore > 1
Stage 2. Percentage of patients with clinical remission | at Week 52
  Clinical remission is defined for a participant to satisfy the following two response thresholds simultaneously: average daily LSF subscore of ≤ 3 as assessed on the CDAI LSF item AND average daily AP subscore of ≤ 1 as assessed on the CDAI AP item (measured by PRO questrionare)
Stage 2: Percentage of patients with CS-free endoscopic remission | at Week 52
  Percentage of patients achieving Endoscopic remission and are CS-free where endoscopic remission is defined as : - SES-CD total score of 0-2, OR - SES-CD total score of ≤ 4 and at least 2 point reduction from Baseline with no subscore > 1
Stage 2. Percentage of patients with CS-free clinical remission | at Week 52
  Percentage of patients achieving CS-free average daily LSF subscore of ≤ 3 as assessed on the CDAI LSF item AND average daily AP subscore of ≤ 1 as assessed on the CDAI AP item
Stage 2: Percentage of patients with CS-free endoscopic remission | at Week 52
  For participants taking CS at Baseline, percentage of patients achieving CS-free endoscopic remission
Stage 2: Percentage of patients with CS-free clinical remission | at Week 52
  For participants taking CS at Baseline, percentage of patients achieving CS-free clinical remission
Stage 2. Percentage of patients with endoscopic response | at Week 12
  Endoscopic response is described as minimum of 50% decrease from Baseline in SES-CD total score
Stage 2. Percentage of patients with clinical remission | at Week 12
  Clinical remission is defined for a participant to satisfy the following two response thresholds simultaneously: average daily LSF subscore of ≤ 3 as assessed on the CDAI LSF item AND average daily AP subscore of ≤ 1 as assessed on the CDAI AP item (measured by PRO questrionare)
Stage 2. Percentage of patients with endoscopic response and endoscopic remission | Endoscopic response at Week 12, endoscopic remission at Week 52
  Endoscopic response is defined as minimum of 50% decrease from Baseline in SES-CD total score Endoscopic remission: - SES-CD total score of 0-2, OR - SES-CD total score of ≤ 4 and at least 2 point reduction from Baseline with no subscore > 1
Stage 2. Percentage of patients with clinical remission | at both Week 12 and Week 52
  Clinical remission is defined for a participant to satisfy the following two response thresholds simultaneously: average daily LSF subscore of ≤ 3 as assessed on the CDAI LSF item AND average daily AP subscore of ≤ 1 as assessed on the CDAI AP item (measured by PRO questionnaire)
Stage 2. Percentage of patients achieving CS-free endoscopic response | at Week 52
  Endoscopic response is described as minimum of 50% decrease from Baseline in SES-CD total score
Stage 2. Percentage of patients with clinical remission | at Week 52
  Percentage of patients achieving CS-free clinical remission Clinical remission is defined for a participant to satisfy the following two response thresholds simultaneously: average daily LSF subscore of ≤ 3 as assessed on the CDAI LSF item AND average daily AP subscore of ≤ 1 as assessed on the CDAI AP item.(measured by PRO questionnaire)
Stage 2. Serum concentration of brazikumab | Through Week 68
  Pharmacokinetics: concentration of brazikumab in serum
Stage 2. Incidence of anti-drug antibodies | Through Week 68
  Immunogenicity: incidence of brazikumab anti-drug antibodies in blood serum
Stage 2. Exposure-response | Through Week 68
  Derive exposure response model linking primary endpoint to metrics of model predicted individual brazikumab exposures
Stage 2. Number and percentage of patients with adverse events | Through Week 68
  Number and percentage of patients with reported adverse events
Stage 2. Percentage of patients with potentially clinically significant changes in laboratory values | Through Week 68
  Percentage of patients with clinically significant changes in hematology, clinical chemistry, urinalysis.
Stage 2. Percentage of patients with potentially clinically significant changes in vital signs | Through Week 68
  Percentage of patients with potentially clinically significant changes in systolic, diastolic pulse rate
Stage 2. Percentage of patients with potentially clinically significant changes in physical exams | Through Week 68
  Percentage of patients with potentially clinically significant changes in full physical exams
Stage 2. Percentage of patients with potentially clinically significant changes in ECGs | Through Week 68
  Percentage of patients with potentially clinically significant changes in 12-lead ECG recordings

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Bohannon, Study Director — AstraZeneca
Locations (89):
- United States (34):
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Lancaster, California
  - Research Site, Lincoln, California
  - Research Site, Poway, California
  - Research Site, San Diego, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Boca Raton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Naples, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Oak Lawn, Illinois
  - Research Site, Brownsburg, Indiana
  - Research Site, Chesterfield, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Morehead City, North Carolina
  - Research Site, Beachwood, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Uniontown, Pennsylvania
  - Research Site, Carrollton, Texas
  - Research Site, Houston, Texas
  - Research Site, McAllen, Texas
  - Research Site, Pflugerville, Texas
  - Research Site, Stafford, Texas
  - Research Site, North Chesterfield, Virginia
  - Research Site, Spokane, Washington
- Canada (2):
  - Research Site, New Westminster, British Columbia
  - Research Site, Chicoutimi, Quebec
- Czechia (4):
  - Research Site, České Budějovice
  - Research Site, Hořovice
  - Research Site, Hradec Králové
  - Research Site, Olomouc
- Germany (7):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Kiel
  - Research Site, Minden
  - Research Site, Remscheid
  - Research Site, Ulm
- Research Site, Budapest, Hungary
- India (4):
  - Research Site, Bangalore
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Surat
- Israel (3):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
- Italy (2):
  - Research Site, Milan
  - Research Site, Padua
- Poland (10):
  - Research Site, Bydgoszcz
  - Research Site, Chojnice
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Sopot
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zamość
- Russia (3):
  - Research Site, Aramil
  - Research Site, Moscow
  - Research Site, Perm
- Slovakia (3):
  - Research Site, Banská Bystrica
  - Research Site, Košice
  - Research Site, Nitra
- South Africa (3):
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Plumstead
- South Korea (3):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seoul
- Spain (3):
  - Research Site, Madrid
  - Research Site, Pontevedra
  - Research Site, Valencia
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Ukraine (2):
  - Research Site, Kharkiv
  - Research Site, Kyiv
- United Kingdom (2):
  - Research Site, Coventry
  - Research Site, West Bromwich

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home